CLINICAL TRIAL: NCT04105179
Title: Do TKA Implant Designs Affect Muscle Mass Change and Muscle Activity During Activities of Daily Living as Well as the Patient Immunological Response
Brief Title: How TKA Implants Affect Muscle Quality and Activity During Daily Living and Immunological Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: University of Ottawa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20180532
Record Dates: First submitted 2018-09-13; First posted 2019-09-26 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Osteoarthritis, Knee; Inflammation Knees
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Implant Groups (Experimental): Group will receive the Smith & Nephew Journey II knee implant or the Zimmer NexGen LPS-Flex knee implant
  Interventions: Device: Zimmer NexGen LPS-Flex; Device: Smith & Nephew Journey II
- Healthy Control Group (No Intervention): Control group that will not be undergoing a total knee arthroplasty

INTERVENTIONS:
Device: Zimmer NexGen LPS-Flex — Patients will be randomly assigned to 1 of 2 devices
  Arms: Implant Groups
Device: Smith & Nephew Journey II — Patients will be randomly assigned to 1 of 2 devices
  Arms: Implant Groups

SUMMARY:
This study compares two total knee replacement implants to asses muscle function and quality, and the immune response to the implants. 30 patients will receive the Smith and Nephew Journey II implant, while 30 patients will receive the Zimmer NexGen LPS-flex implant. 15 healthy controls will also be recruited and compared.

DETAILED DESCRIPTION:
Patients will undergo biomechanics testing while they complete sit-to-stand, stand-to-sit, lateral step down, level walking, and single leg balance tasks up to 1 month before surgery, and 6 and 12 months after surgery. They will also undergo MRI imaging up to 1 month before surgery and 12 months after surgery to assess muscle quality. A secondary outcome will also be to analyze the immunological response in the patients who received femoral components made of oxidized zirconium versus contemporary components made of cobalt chrome. Fifteen healthy controls will also participate in the study and will undergo the biomechanical, MRI and blood draws at a single visit.

ELIGIBILITY:
Inclusion Criteria:

* The participants receiving a knee implant must requiring a total knee replacement

Exclusion Criteria:

* Any degenerative conditions (other than osteoarthritis at the affected knee) impacting joints of the lower extremities
* bilateral knee replacements
* previous joint replacement at the affected knee
* any other past or present conditions that may impact gait
* any active infection and any diagnosed conditions that may affect the local and systemic immune response (e.g., rheumatoid arthritis, HIV infection, lupus, pregnancy, and thrombocytosis)
* BMI and waist circumference (WC) will be another exclusion criterion since both BMI and WC are associated with health problems and gait abnormalities. Any patient with both BMI > 35 kg/m2 and a WC > 102 cm in men or > 88 cm in women will be excluded from the study.

Healthy Controls Inclusion

* controls must not suffer from lower extremity injuries or joint conditions that might alter gait dynamics Exclusion
* BMI and waist circumference (WC) will be another exclusion criterion since both BMI and WC are associated with health problems and gait abnormalities. Any patient with both BMI > 35 kg/m2 and a WC > 102 cm in men or > 88 cm in women will be excluded from the study

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2019-04-29 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline knee extension moment at 6 and 12 months during gait | Baseline (within 1 month of surgery), 6 months post-surgery, and 12 months post-surgery; and versus healthy controls
  Peak knee extension moment will be measured by combining three-dimensional images of movement with time, the knee extension will be calculated in degrees while the participant walks at their normal walking speed.
Change from baseline muscle quality assessed via MRI at 12 months | Baseline (within 1 month of surgery), 12 months post-surgery; and versus healthy controls
  Proton density fat fraction of the quadriceps and hamstrings muscles will be measured via MRI
Change from baseline quadriceps muscle activation at 6 and 12 months during gait | Baseline (within 1 month of surgery), 6 months post-surgery, and 12 months post-surgery; and versus healthy controls
  Peak muscle activation of the quadriceps muscle will be measured with electromyography while the participant walks at their normal walking speed

SECONDARY OUTCOMES:
Change in trace metal concentrations from baseline, 12 months, and 24 months | Baseline (within 1 month of surgery), 12 months post-surgery, 24 months post-surgery; and versus healthy controls
  Peripheral blood will be collected prior to surgery and at 12 months post-surgery; for symptomatic patients, a third blood draw will occur at 24 months post-surgery. Concentrations of cobalt, chromium, and Nickle will be measured by inductively coupled plasma-mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Lamontagne, PhD, Principal Investigator — University of Ottawa; Isabelle Catelas, PhD, PEng, Principal Investigator — University of Ottawa
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR